CLINICAL TRIAL: NCT05682924
Title: Condition Vasoregulation Function Endothelium in Patients With Chronic Myeloid Leukemia (CML) Getting Tyrosine Kinase Inhibitor (TKI) II Generation Bosutinib
Brief Title: Condition Vasoregulation Function Endothelium in Patients With CML Getting TKI II Generation Bosutinib
Status: Recruiting | Type: Observational
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20221112
Record Dates: First submitted 2022-12-14; First posted 2023-01-12 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Chronic Myeloid Leukaemia
Keywords: chronic myeloid leukaemia; tyrosine kinase inhibitor; endothelium; endothelial dysfunction; bosutinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group: 35 patients with ph-positive chronic myeloid leukemia in the chronic phase, aged 40 to 60 years, receiving bosutinib at a dose of 500 mg / day
  Interventions: Diagnostic Test: taking blood for the study of biochemical parameters and the study of microcirculation using the method of laser Doppler flowmetry
- Comparison group: 35 patients with ph-positive chronic myeloid leukemia in the chronic phase, aged 40 to 60 years, receiving nilotinib at a dose of 800 mg / day
  Interventions: Diagnostic Test: taking blood for the study of biochemical parameters and the study of microcirculation using the method of laser Doppler flowmetry
- Control group: 35 patients with ph-positive chronic myeloid leukemia in the chronic phase, aged 40 to 60 years, receiving imatinib at a dose of 600 mg / day
  Interventions: Diagnostic Test: taking blood for the study of biochemical parameters and the study of microcirculation using the method of laser Doppler flowmetry

INTERVENTIONS:
Diagnostic Test: taking blood for the study of biochemical parameters and the study of microcirculation using the method of laser Doppler flowmetry — In the study, blood will be taken from patients with chronic myelogenous leukemia in the chronic phase to determine biochemical parameters (endothelin-1, homocysteine, VEGF (vascular endothelial growth factor)), as well as a study of microcirculation in these groups of patients using the method of laser Doppler flowmetry, to study the function of the endothelium.

SUMMARY:
The study will study the state of the endothelium in patients with chronic myeloid leukemia during therapy with the II generation tyrosine kinase inhibitor bosutinib. Patients will be divided into groups receiving nilotinib 800mg/day, bosutinib 500mg/day, and imatinib 600mg/day. A comprehensive examination of patients will be carried out, including a clinical examination, a study of biochemical markers of endothelial damage and the functional state of the vascular wall. An algorithm will be developed for assessing the state of endothelial function in patients with ph-positive chronic myeloid leukemia in the chronic phase when using the second-generation tyrosine kinase inhibitor bosutinib.

DETAILED DESCRIPTION:
Purpose: To assess the state of endothelial vasoregulatory function in patients with chronic myelogenous leukemia receiving the II generation tyrosine kinase inhibitor bosutinib as a second line of therapy based on a comprehensive assessment of biochemical markers of endothelial damage and the results of laser Doppler flowmetry.

Description of the Protocol: At the first stage, study groups will be formed. The study groups will consist of 70 patients with ph-positive chronic myeloid leukemia in the chronic phase, aged 40 to 60 years, receiving nilotinib at a dose of 800 mg / day. (35 people) and bosutinib at a dose of 500 mg/day. (35 people) matched by sex and age. The control group will consist of 35 patients matched by gender and age with ph-positive chronic myeloid leukemia in the chronic phase, aged 40 to 60 years, receiving imatinib at a dose of 600 mg/day. (35 people).

At the second stage, it is planned to conduct a comprehensive examination of patients, including a clinical examination, a study of biochemical markers of endothelial damage and the functional state of the vascular wall.

At the third stage, the relationship between the results of laboratory methods for assessing endothelial function and dynamic parameters of microcirculation, determined by laser Doppler flowmetry in patients with ph-positive chronic myeloid leukemia in the chronic phase, receiving therapy with the II generation tyrosine kinase inhibitor bosutinib, will be analyzed.

At the fourth stage, it is planned to develop an algorithm for assessing the state of endothelial function in patients with ph-positive chronic myelogenous leukemia in the chronic phase using the second generation tyrosine kinase inhibitor bosutinib.

Scientific novelty

1. For the first time, an assessment of the state of endothelial function will be given on the basis of a comprehensive study using the Doppler flowmetry method and the determination of biochemical indicators of endothelial damage in patients with ph-positive chronic myeloid leukemia in the chronic phase while taking the II generation tyrosine kinase inhibitor bosutinib.
2. For the first time, an algorithm will be proposed for diagnosing the state of endothelial function in patients with ph-positive chronic myeloid leukemia in the chronic phase when using therapy with the II generation tyrosine kinase inhibitor bosutinib, based on the use of a multifactorial method of mathematical modeling.

Practical significance Indicators will be determined that reflect the state of the vasoregulatory function of the endothelium in patients with ph-positive chronic myeloid leukemia in the chronic phase when using therapy with II generation tyrosine kinase inhibitors bosutinib.

Taking into account the identified changes, an algorithm will be developed for assessing the state of endothelial function in patients with ph-positive chronic myeloid leukemia in the chronic phase when using the second-generation tyrosine kinase inhibitor bosutinib.

Expected results Based on a comprehensive analysis of indicators of endothelial vasoregulatory function, including biochemical parameters and an assessment of the information content of the laser Doppler flowmetry method, an algorithm for assessing the state of endothelial function in patients with ph-positive chronic myeloid leukemia in the chronic phase against the background of taking the II generation tyrosine kinase inhibitor bosutinib will be developed.

ELIGIBILITY:
Inclusion Criteria:

* patients with ph-positive chronic myeloid leukemia in the chronic phase before treatment and taking tyrosine kinase inhibitors of I and II generations (imatinib, nilotinib, bosutinib);
* availability of informed consent of the patient to participate in the study.

Exclusion Criteria:

* history of acute cerebrovascular accident;
* previous myocardial infarction in anamnesis;
* the presence of diabetes mellitus type I and II;
* the presence of chronic kidney disease C1-C5 stages;
* the presence of coronary heart disease with its clinical manifestations (II-IV functional class);
* the presence of hypertension III degree;
* the presence of atherosclerotic lesions of peripheral arteries according to the color duplex sonography data of the arteries of the upper and lower extremities;
* atrial fibrillation and flutter;
* the presence of other oncological diseases;
* inflammatory diseases in the acute stage;
* the presence of mutations, in which the appointment of tyrosine kinase inhibitors of the I or II generation is not indicated (resistance to tyrosine kinase inhibitors drugs)
* refusal of the patient from examination.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with ph-positive chronic myeloid leukemia in the chronic phase, aged 40 to 60 years, who meet the inclusion/exclusion criteria, receiving therapy with the tyrosine kinase inhibitors II generation bosutinib, nilotinib, and the tyrosine kinase inhibitors I generation imatinib.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of type of microcirculation. | 3 months
  Type of microcirculation (normal, hyperemic, spastic, congestive) according to the LAKK-OP apparatus

SECONDARY OUTCOMES:
Confirmation or exclusion of endothelial dysfunction. | during inclusion
  Biochemical marker - Human Endothelin 1 (ET-1), fmol/ml
Confirmation or exclusion of endothelial dysfunction. | 3 months
  Biochemical marker - VEGF (vascular endothelial growth factor), pg/ml
Confirmation or exclusion of endothelial dysfunction. | 6 months
  Biochemical marker - Homocysteine, µmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Cherenova, Principal Investigator — Samara State Medical University
Locations (2):
- Russia (2):
  - National Medical Research Centre for Hematology, Moscow
  - Samara State Medical University, Samara

IPD SHARING:
Plan to Share IPD: Undecided